CLINICAL TRIAL: NCT04068324
Title: Comparison of Postoperative Recovery After Preoperative Carbohydrate Loading With Standard Fasting in Pediatric Patients Undergoing Nuss Operation
Brief Title: Postoperative Recovery Quality According to Preoperative Fasting Time in Pediatric Patients Undergoing Nuss Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jung Min Koo (Other)
Responsible Party: Sponsor-Investigator, Jung Min Koo, Principal Investigator, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: KC19ENSI0335
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 8 hours fasting group (No Intervention): Routine preoperative fasting group undergoes 8 hours of fasting before the operation.
- Clear liquid group (Experimental): 30 pediatric patients drink 3ml/kg 1 hour before the surgery. Although "clear liquid" suggests any drinks that do not contain any solid ingredients, but in this study we define "clear liquid" as water.
  Interventions: Dietary Supplement: New Care No Nil Per Os
- Carbohydrate containing liquid group (Experimental): Other 30 pediatric patients drink 3ml/kg of carbohydrate containing fluid 1 hour before the surgery. The product name we have is "NoNPO" from NewCare (South Korean company). This fluid does not contain any solid ingredients, so consuming the fluid does not exceed Nil per Os time needed before the surgery.
  Interventions: Dietary Supplement: New Care No Nil Per Os

INTERVENTIONS:
Dietary Supplement: New Care No Nil Per Os — The product name "NoNPO" is from South Korean company "Well life." It contains carbohydrate and is frequently used in preoperative fasting patients in order to alleviate patients' discomfort resulting from empty stomach and thirst. It is also known to decrease insulin resistant.
  Arms: Carbohydrate containing liquid group; Clear liquid group

SUMMARY:
Preoperative fasting is intended to lower the amount of gastric contents in order to decrease the incidence of aspiration associated with endotracheal intubation. However, recent studies show that longer fasting time does not reduce aspiration associated complications. Especially in pediatric patients, long fasting time increases patients' unpleasantness and therefore increases postoperative recovery quality. It also induces hypoglycemia. In many studies, ingesting clear liquids 2 hours up to general anesthesia decreases gastric contents and therefore the incidence of aspiration pneumonia, postoperative nausea and vomiting. Therefore anesthesiologist associations in the US and Europe recommend to drink small amount of clear liquid (water) up to 2 hours before the surgery.

Nuss bar operation, or repair surgery of pectus excavatum is mostly done in pediatric patients. The procedure itself is very painful, requiring paramount amount of analgesics. Use of opioid analgesics increases postoperative nausea and vomiting.

In this study, our aim is to evaluate preoperative fasting time and how preoperative supplement of clear liquid affects the quality of recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients from age 3 to 6
2. Undergoing repair surgery for pectus excavatum
3. American Society of Anesthesiologists class I to III

Exclusion Criteria:

1. Any diseases or past surgical procedures involving gastrointestinal tract
2. Past history of psychiatric diseases
3. On chronic analgesic medication
4. Patients or Patients' caregivers do not agree to attend the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2021-01-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Modified-Yale Preoperative Anxiety Scale | Preoperatively at the surgery waiting room
  MyPas scale measures 4 categories: Activity, Vocalizations, Emotional Expressivity and State of Apprent Arousal. Each category has 1 to 4 scales for activity, emotional expresivity and state of apprent arousal, and 1 to 6 for vocalizations, that each describes the child's anxiety status. The observer collects total score ranging from 4 to 18.
Emergence delirium | 5 Minutes postoperatively at postoperative discharge unit
  "Watcha scale" measures child's postoperative delirium at the recovery center. The total score ranges from 0 to 4. 0 is when the child is asleep, 1 is calm and sedated, 2 is when the child is crying but consolable, 3 is when the child is crying and unconsolable, and 4 is when the child is uncontrollable.
Emergence delirium | 10 Minutes postoperatively at postoperative discharge unit
  "Watcha scale" measures child's postoperative delirium at the recovery center. The total score ranges from 0 to 4. 0 is when the child is asleep, 1 is calm and sedated, 2 is when the child is crying but consolable, 3 is when the child is crying and unconsolable, and 4 is when the child is uncontrollable.
Emergence delirium | 15 Minutes postoperatively at postoperative discharge unit
  "Watcha scale" measures child's postoperative delirium at the recovery center. The total score ranges from 0 to 4. 0 is when the child is asleep, 1 is calm and sedated, 2 is when the child is crying but consolable, 3 is when the child is crying and unconsolable, and 4 is when the child is uncontrollable.
Emergence delirium | 30 Minutes postoperatively at postoperative discharge unit
  "Watcha scale" measures child's postoperative delirium at the recovery center. The total score ranges from 0 to 4. 0 is when the child is asleep, 1 is calm and sedated, 2 is when the child is crying but consolable, 3 is when the child is crying and unconsolable, and 4 is when the child is uncontrollable.
Emergence delirium | 45 Minutes postoperatively at postoperative discharge unit
  "Watcha scale" measures child's postoperative delirium at the recovery center. The total score ranges from 0 to 4. 0 is when the child is asleep, 1 is calm and sedated, 2 is when the child is crying but consolable, 3 is when the child is crying and unconsolable, and 4 is when the child is uncontrollable.
Emergence delirium | 60 Minutes postoperatively
  "Watcha scale" measures child's postoperative delirium at the recovery center. The total score ranges from 0 to 4. 0 is when the child is asleep, 1 is calm and sedated, 2 is when the child is crying but consolable, 3 is when the child is crying and unconsolable, and 4 is when the child is uncontrollable.
Pain Score | 5 minutes postoperatively at postoperative discharge unit
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.
Pain Score | 10 minutes postoperatively at postoperative discharge unit
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.
Pain Score | 15 minutes postoperatively at postoperative discharge unit
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.
Pain Score | 30 minutes postoperatively at postoperative discharge unit
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.

SECONDARY OUTCOMES:
Pain scores | Between 1~6 hours postoperatively
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.
Pain scores | Between 12~24 hours postoperatively
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.
Pain scores | Between 24~48 hours postoperatively
  Face, Legs, Activity, Cry and Consolability score: This is a measurement for pediatric pain. The observer observes the child's face, legs, activity, cry and consolability. The score ranges from 0 to maximum of 8. 0 is when the child is calm without any pain, and 8 being the most painful expression of the child.
Other pro re nata analgesics used, amount and type | Between 1~6 hours postoperatively
  Analgesics applied in the ward according to the child's pain scale or as requested by his or her parents
Other pro re nata analgesics used, amount and type | Between 12~24 hours postoperatively
  Analgesics applied in the ward according to the child's pain scale or as requested by his or her parents
Other pro re nata analgesics used, amount and type | Between 24~48 hours postoperatively
  Analgesics applied in the ward according to the child's pain scale or as requested by his or her parents
Any postoperative side effects | Between 1~6 hours postoperatively
Any postoperative side effects | Between 12~24 hours postoperatively
Any postoperative side effects | Between 24~48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min Koo, MD, Principal Investigator — Seoul St. Mary's Hospital, South Korea
Locations (1):
- Jung Min Koo, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided